CLINICAL TRIAL: NCT03242876
Title: The Effects of Citric and Malic Acid Found in Pomegranate Juice on Glycaemic Response
Brief Title: The Effects of Citric and Malic Acid Found in Pomegranate Juice on Glycaemic Response to White Bread.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Gary Williamson, Prof functional foods, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MEEC 15-044a
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Hyperglycemia, Postprandial
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control meal (Placebo Comparator): Control will be 109 g white bread and 200 mL water. The glycaemic response to the test meal will be compared to the response of the control meal.
  Interventions: Other: Control
- Test meal (Experimental): Test will be 109 g white bread and 200 mL water containing 3.819 g citric acid and 119 mg malic acid adjusted to pH 3.2. The glycaemic response to this meal will be compared to that of the control meal.
  Interventions: Other: Test

INTERVENTIONS:
Other: Control — Control will be 109 g white bread to be consumed together with 200 mL water
  Arms: Control meal
Other: Test — Test will be 109 g white bread to be consumed together with 3.819 g citric acid and 119 mg malic acid dissolved in 200 mL water adjusted to pH 3.2.
  Arms: Test meal

SUMMARY:
Research has shown that diets that give rise to a high glucose response are associated with a number of abnormalities like increased risk of metabolic syndrome. Metabolic syndrome mostly comprises of insulin resistance and glucose intolerance which gives an increased risk of type 2 diabetes. It also gives rise to other conditions like high blood pressure (arterial hypertension), elevated blood insulin levels (hyper-insulinemia), elevated amounts of fat in the liver (fatty hepatosis) and elevated amounts of lipids in the blood (dyslipidemia). After type 2 diabetes become clinically apparent, the risk of cardiovascular disease also rises. Research has also shown that foods/drinks which raise blood glucose levels gradually (low GI) rather than rapidly (high GI) have health benefits which include reducing the risk of metabolic syndrome. Laboratory studies have shown that polyphenols found in fruits, vegetables and plant based foods have a positive effect on carbohydrate metabolism and can lower the blood glucose levels.

Therefore a lower glycemic index diet may have benefits in terms of type two diabetes and heart disease management, and as a method for weight loss. There has been some research into the effects of pomegranate on lowering blood glucose responses both chronically and acutely. Mechanistic evidence suggests that this effect could be down to the organic acids found within pomegranate juice. 16 volunteers were fed 50 g available carbohydrate from white bread (109 g), and either 200 ml water (control) or 200 ml solution (test) containing citric acid (3.8 g) and malic acid (119 mg) the quantities that are found in 200 ml pomegranate juice (Biona) as analysed. Blood glucose was measured at baseline, and at 30 - 60 minute increments over three hours. Glucose curves were plotted, and the area under the curve was calculated and compared between conditions for each participant.

DETAILED DESCRIPTION:
The world health organisation has reported that over 220 million people suffer from diabetes worldwide and that by the year 2030, this number will be doubled. The WHO also reports that in 2004, about 3.4 million people died from high blood sugar. About 90% of all diabetes cases is due to type II diabetes. Type 2 diabetes is largely due to overweight and lack of physical activity characterised by high glucose levels (hyperglycaemia).

In the human diet, the source of blood glucose is carbohydrates. Dietary carbohydrate is important to maintain glycaemic homeostasis and provides the most of the energy in the diets of most people. The control of blood glucose is a hormonal process and it is very important to human physiology. Hormonal processes involve the release of insulin from the β- cells of the pancreatic cells which stimulates the uptake of glucose after a meal, to other tissues either for utilisation (glycolysis) or to be stored in the liver as glycogen (glycogenesis). When blood glucose falls below normal, glucagon is secreted from the pancreatic α-cells and it promotes liver glucose production by inducing the generation of glucose from non-carbohydrate substrates such as amino and fatty acids (gluconeogenesis) and the generation of glucose from glycogen (glycogenolysis).

When the glucose homeostasis hormonal control fails, it entails high blood glucose levels (postprandial hyperglycaemia) which can lead to metabolic syndrome which includes obesity, impaired glucose tolerance (IGT), hypertension and dyslipidemia. Disturbance of glucose homeostasis can also lead to other symptoms such as inflammation and oxidative stress at the whole body level as well as disturbances of the functionality in several organs as well as diabetes. Therefore, as much as carbohydrates are required in the human body as a major source of energy, too much in the diet can have adverse health effects especially the one with high glycaemic effect.

The proposed mechanism adapted from Aston, 2006 of how carbohydrates may affect human health is that when there is a continual presence of high glycaemic index foods in the diet, this gives rise to postprandial glucose rise as well as high insulin demand to act on the high blood glucose levels in the blood. Postprandial glucose rise and high insulin demand may lead to insulin resistance which is the major component of metabolic syndrome. High insulin demand may also lead to β-cell failure which may also result in hyperglycaemia which is also a cause of insulin resistance. Insulin resistance and hyperglycaemia are risk factors for metabolic syndrome and diabetes type 2.

Scientific evidence suggest that postprandial hyperglycaemia in humans has a major role to play in health priorities like type 2 diabetes and blood glucose control. It has been reported that about 90% of all diabetes cases consist of type 2 diabetes. Apart from type I and type 2 diabetes, there are other related conditions which include pre-diabetes (impaired glucose tolerance (IGT) and impaired fasting glucose (IFG) as well as metabolic syndrome (obesity, hypertension and insulin resistance). It has been reported that pre-diabetes and metabolic syndrome increases the risk of developing cardiovascular disease and diabetes mellitus. The glycaemic index was originally proposed with the aim of managing diabetes. However, recent studies have shown that the GI has potential in the prevention of type 2 diabetes as well as in the treatment of metabolic syndrome. Research has shown that high GI diets are associated with increased risk of developing type 2 diabetes. More research has shown that high GI diet is associated with a number of abnormalities like increased metabolic syndrome and insulin resistance. In the same way, a low GI diet is said to improve insulin sensitivity but more research is needed to support this. A few studies have shown this to be the case. However it was observed that it was difficult to know whether this was as a result of improved insulin sensitivity, or improved insulin secretion or due to reduced rate of glucose absorption.

Potential solution having anything in the diet that can either slow down the digestion and absorption of carbohydrates can help reduce the risk. Among others, two potential solutions are that of consumption of low glycaemic index foods or having ingredients in the diet that can reduce the glycaemic index of foods as well as postprandial blood glucose levels. The presence of inhibiting components in the diet that can reduce postprandial glucose can also be a solution to reducing the risk. Drugs like acarbose are currently used in some countries for the management of type 2 diabetes which act by inhibiting carbohydrate digestive enzymes. However, the use of acarbose has side effects such as nausea, flatulence and diarrhoea. It has been reported that polyphenols also have the potential to inhibit the rise in blood glucose by hindering the rapid absorption of glucose.

A recent review has reported that research using animal models as well as a limited number of human studies, have shown that polyphenols and polyphenol rich foods or beverages have the potential to affect postprandial glycaemic responses and fasting glycaemia as well as an improvement of acute insulin secretion and sensitivity. Other possible mechanisms as reported in the review include pancreatic β- cells stimulation to secrete insulin as well as activation of insulin receptors, modulation of the release of glucose from the liver as well as of intracellular signalling pathways and gene expression.

Another recent review concluded that it is very possible that the effects of polyphenols in the diet will affect glycaemic index of foods as well as postprandial glucose responses in humans. The two mechanisms highlighted by which this can be achieved being the inhibition of sugar metabolising enzymes as well as transporters. This potential action of polyphenols can thus be compared to that of acarbose which acts by the same mechanism and research in chronic intervention studies has shown that it reduces diabetes risk.

This study was carried out as a parallel control to another study which looked at the effects of polyphenols found in pomegranate juice. The aim was to determine the effects of the acids found in the pomegranate juice on glycaemic response to bread.

ELIGIBILITY:
Inclusion Criteria:

* Measured on first visit: Fasting glucose (blood glucose level before breakfast) 3.9 -5.9 mmol/L
* Apparently healthy
* Not diabetic
* Not on long term prescribed medication (except contraceptives)
* Not pregnant or lactating
* Not on special diet (for losing weight or fruit extract supplements)
* Aged 18-75

Exclusion Criteria:

* Measured fasting plasma glucose >5.9 mmol/L
* Not healthy
* Diabetic
* Pregnant or lactating
* On special diet (for losing weight)
* On long term prescribed medication
* Smoker
* Diabetic

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Incremental area under the glucose curve | 1 year
  The incremental area under the glucose curve after consumption of the test meal will be compared to that obtained after the control meal

CONTACTS AND LOCATIONS:
Overall Officials: Gary Williamson, PhD, Study Chair — University of Leeds; Hilda Nyambe, PhD, Principal Investigator — University of Leeds
Locations (1):
- School of Food Science and Nutrition, University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kerimi A, Nyambe-Silavwe H, Gauer JS, Tomas-Barberan FA, Williamson G. Pomegranate juice, but not an extract, confers a lower glycemic response on a high-glycemic index food: randomized, crossover, controlled trials in healthy subjects. Am J Clin Nutr. 2017 Dec;106(6):1384-1393. doi: 10.3945/ajcn.117.161968. Epub 2017 Oct 11. PMID 29021286